CLINICAL TRIAL: NCT04330937
Title: Clinical Trial on the Effectiveness of Citrolive® to Decrease Oxidation of Low Density Lipoproteins
Brief Title: Clinical Trial on the Effectiveness of Citrolive
Acronym: CITROXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-0008
Record Dates: First submitted 2019-10-16; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): volunteers consume 1 capsule per day for 3 months. (500 mg citrolive).
  Interventions: Dietary Supplement: dietetics
- control group Placebo (sucrose) (Placebo Comparator): volunteers consume 1 capsule per day for 3 months. (saccharose).
  Interventions: Dietary Supplement: dietetics

INTERVENTIONS:
Dietary Supplement: dietetics — 90 days of consumption

SUMMARY:
The clinical trial consists in checking the antioxidant effect of citrolive on low density cholesterol.

DETAILED DESCRIPTION:
The clinical trial consists in checking the antioxidant effect of citrolive on low density cholesterol. To do this, volunteers consume the product under study or placebo for three months.

Tests will be performed before and after ingestion of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Not belonging to the group of individuals considered as priorities by the Third Joint Task Force for the prevention of cardiovascular diseases due to high risk.
2. Present total cholesterol figures greater than 200 milligrams / deciliter and / or low density cholesterol figures greater than 130 milligrams / deciliter so that after applying the cardiovascular risk table (SCORE) they present a current risk of less than 5% of suffer an ischemic event in a period of 10 years, being without pharmacological treatment.
3. Present several cardiovascular risk factors with cholesterolemia figures close to 200 milligrams / deciliters and / or low density cholesterol figures close to 130 milligrams / deciliters.

Exclusion Criteria:

1. chronic or terminal illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | The change in systolic and diastolic blood pressure is observed after three months of intake of the product under investigation
  The systolic and diastolic blood pressure was measured with an OMRON oscilimétrilo sphygmomanometer
Biochemistry and blood count | The change is observed after three months of intake of the product under investigation
  the hematological profile is analyzed with the Horiba ABX Oentra 80 analyzer. Biochemical profile with the ILAB 600 analyzer

SECONDARY OUTCOMES:
Weight | The change is observed after three months of intake of the product under investigation
  Measured in Kg.
Height | The change is observed after three months of intake of the product under investigation
  Measured in cm.
BMI | The change is observed after three months of intake of the product under investigation
  Weight and height are combined for BMI report in kg / m ^ 2
Perimeters | The change is observed after three months of intake of the product under investigation
  Measured in cm. Waist, hip, waist / hip index, relaxed biceps, contracted biceps, medial thigh, twin or calf.
  Folds (mm) (tricipítal, subscapular, suprailiac anterior or supraspinal, abdominal, quadricipital or thigh, leg or calf medial, bicipital, iliocrestal).
  Diameters (cm) (radiocubital or wrist biestiloid, humeral or elbow bicpicondiolo, femoral or knee bicondiol).
Folds | The change is observed after three months of intake of the product under investigation
  Measured in mm. Tricipítal, subscapular, suprailiac anterior or supraspinal, abdominal, quadricipital or thigh, leg or calf medial, bicipital, iliocrestal.
  Diameters (cm) (radiocubital or wrist biestiloid, humeral or elbow bicpicondiolo, femoral or knee bicondiol).
Diameters | The change is observed after three months of intake of the product under investigation
  Measured in cm. Radiocubital or wrist biestiloid, humeral or elbow bicpicondiolo, femoral or knee bicondiol.
Nutritional record | Measurements are made at the beginning and after 90 days of product consumption.
  Volunteers record dietary intake for three days in a notebook. They will describe the amount of food they consume in grams in order to assess changes in intake during the clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain